CLINICAL TRIAL: NCT00423891
Title: Evaluation of the Pharmacokinetics, Safety, Tolerability and Efficacy of Entecavir (ETV) in Pediatric Subjects With Chronic Hepatitis B Virus (HBV) Infection Who Are HBeAg-Positive
Brief Title: A Study of Entecavir in Pediatric Patients With Chronic Hepatitis B Virus (HBV)-Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI463-028
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1: Entecavir (Experimental)
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — Tablets / Oral Solution, Oral, Naïve: 0.015 mg/kg up to 0.5 mg; Experienced: 0.030 mg/kg up to 1 mg, once daily, 48 - 120 weeks depending on response
  Other Names: Baraclude; BMS-200475

SUMMARY:
The purpose of this clinical study is to determine the appropriate doses of entecavir to use in children and adolescents. Safety, tolerability and efficacy will also be studied

ELIGIBILITY:
Inclusion Criteria:

* 2-18 years of age
* Group A: Lamivudine naive (<1 week of Lamivudine) and not within 24 weeks of screening; Group B: Lamivudine experienced (> 12 weeks of Lamivudine); Group C: nucleoside/nucleotide experienced (> 12 weeks of nucleoside/tide therapy) added as a country-specific protocol amendment (not all sites had Group C).
* HBV Deoxyribonucleic acid (DNA) ≥ 100000 copies/mL; ≥ 10000 copies for nucleoside/nucleotide experienced (Group C)
* Detectable Hepatitis B surface antigen (HBsAg) for 24 weeks prior to screening
* Hepatitis B e antigen (HBeAg) positive
* Compensated liver and renal function
* Elevated alanine aminotransferase (ALT) at screening and during the 24 weeks prior to screening (for Groups A and B)

Exclusion Criteria:

* Coinfection with Human immunodeficiency virus (HIV), Hepatitis C virus (HCV), Hepatitis D Virus (HDV)
* Children who were breastfed while their mother received Lamivudine, or children whose mothers received Lamivudine during pregnancy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2007-06-30 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2017-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- United States (9):
  - University of California, San Francisco, San Francisco, California
  - Connecticut Children'S Medical Center, Hartford, Connecticut
  - University Of Florida, Gainesville, Florida
  - Johns Hopkins School Of Medicine, Baltimore, Maryland
  - Boston Childrens Hospital, Boston, Massachusetts
  - Mount Sinai School Of Medicine, New York, New York
  - Children'S Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University Of Texas Southwestern Medical Center, Dallas, Texas
- Local Institution, Buenos Aires, Argentina
- Local Institution, Brussels, Belgium
- Brazil (2):
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Sco Paulo, São Paulo
- Local Institution, Toronto, Ontario, Canada
- Local Institution, Seoul, South Korea
- Local Institution, Taipei, Taiwan
- United Kingdom (2):
  - Local Institution, London, Greater London
  - Local Institution, Birmingham, West Midlands

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 64 enrolled. 48 treated. Participants received a minimum of 48 weeks study drug but depending on response to drug, could remain on treatment for up to a total of 120 weeks. Participants were to receive post dosing follow up after last dose, for a total of 5 years on-study (on and off study drug).
Groups:
- Lamivudine (LVD)-Naive (Group A): Participants with less than (<) 1 week of prior LVD therapy and with no LVD therapy within 24 weeks prior to enrollment were included in Group A. Prior to Pharmacokinetic (PK) assessment, Cohort 1 (age ≥ 2 years to ≤ 6 years) and Cohort 2 (>6 years to ≤ 12 years) received ETV oral solution, 0.015 mg/kg up to 0.5 mg, once a day (QD) and Cohort 3 (age >12 years to ≤18 years) received ETV oral solution, 0.015 mg/kg up to 0.5 mg, or ETV tablets, 0.5 mg, QD. Following PK analysis, those who met the specified dosing requirements (at least 0.5 mg/day) and could tolerate swallowing ETV tablets were allowed to choose either formulation. Entecavir (ETV) was administered for a maximum of 120 weeks.
- Lamivudine (LVD)-Experienced (Group B): Participants with greater than (>) 12 weeks of prior LVD therapy were included in Group B. Prior to PK assessment, Cohort 1 (age ≥ 2 years to ≤ 6 years) and Cohort 2 (> 6 years to ≤ 12 years) received ETV oral solution, 0.030 mg/kg up to 1.0 mg, QD and Cohort 3 (age >12 years to ≤18 years) received ETV oral solution, 0.030 mg/kg up to 1.0 mg, or ETV tablets, 1.0 mg QD. Following PK analysis, those who met the specified dosing requirements (at least 1.0 mg/day) and could tolerate swallowing ETV tablets were allowed to choose either formulation. Entecavir (ETV) was administered for a maximum of 120 weeks.
- Nucleoside/Tide Analog (NA) - Experienced (Group C): Participants who failed previous treatment with any non-ETV nucleoside/tide analog (NA) were included in Group C, starting in 2011. PK assessment was optional to participants in Group C. All participants received ETV oral solution, 0.030 mg/kg up to 1.0 mg, or ETV tablets, 1.0 mg, QD. Participants who met the specified dosing requirements (at least 1.0 mg/day for NA-experienced participants) and could tolerate swallowing ETV tablets were allowed to choose either formulation. ETV was administered for a maximum of 120 weeks.
Period: Enrolled
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Started | 35 | 21 | 8
Completed | 24 | 19 | 5
Not Completed | 11 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — No longer met criteria | 11 | 2 | 1
Period: Treatment
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Started | 24 | 19 | 5
Completed | 22 | 19 | 5
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Post-Dosing Follow Up
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Started | 22 | 18 | 5
Completed | 20 | 15 | 3
Not Completed | 2 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 2
Not completed — Lost to Follow-up | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C) | Total
Number analyzed (Participants) | 24 | 19 | 5 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (5.41) | 11.0 (4.42) | 8.8 (5.02) | 9.9 (4.98)
Age, Customized [Number; unit: participants]
  ≥ 2 years to ≤ 6 years | 7 | 3 | 2 | 12
  >6 years to ≤ 12 years | 9 | 7 | 2 | 18
  >12 years to ≤18 years | 8 | 9 | 1 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 2 | 23
  Male | 10 | 12 | 3 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 17 | 10 | 5 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 2 | 0 | 2
  White | 5 | 6 | 0 | 11
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 1 | 16
  Taiwan | 3 | 0 | 0 | 3
  Canada | 1 | 0 | 0 | 1
  Argentina | 3 | 0 | 0 | 3
  Belgium | 1 | 1 | 0 | 2
  Brazil | 1 | 3 | 0 | 4
  United Kingdom | 2 | 1 | 0 | 3
  Korea, Republic of | 3 | 9 | 4 | 16
Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) [Mean (Standard Deviation); unit: log10 IU/mL] — Hepatitis B virus DNA by polymerase chain reaction (PCR) was measured using the Roche COBAS TaqMan - high pure system (HPS) assay and was reported in international units per milliliter (IU/mL).
  log10 IU/mL | 7.92 (0.864) | 7.74 (0.856) | 7.96 (0.238) | 7.85 (0.812)
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: U/L] — The normal range for serum ALT as established by the study's central laboratory was 5 - 45 units per liter (U/L). The inclusion criteria for Groups A and B was >= 2 X ULN to <= 10 X ULN, while only the upper range applied to Group C (<= 10 X ULN).
  U/L | 142.8 (85.18) | 125.7 (67.96) | 44.6 (22.96) | 125.8 (78.83)

OUTCOME MEASURES:

1. Secondary Outcome: Mean Maximum Observed Plasma Concentration (Cmax) and Mean Trough Observed Plasma Concentration (Cmin) of Entecavir in LVD-naive and LVD-experienced Participants, by Age Cohort
Description: Cmax and Cmin were derived from plasma concentration of ETV versus time and measured in nanograms per milliliters (ng/mL). Blood samples were obtained before study drug administration and at 0.5, 1, 2, 4, 8, and 24 hours after study drug administration on Day 14 (+/- 4 days) for the PK assessment. Plasma samples were analyzed for ETV with a validated method using liquid chromatography-tandem mass spectrometry detection. Note: PK parameters were summarized for only Groups A and B. PK assessment was optional for Group C participants (NA-experienced participants who were included with the September 2011 country-specific protocol amendment). No Group C participants chose to participate in the PK assessment.
Time Frame: Day 14
Population: Participants in Groups A and B who received study drug and had PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B)
Number analyzed (Participants) | 24 | 19
ng/mL
  Cmax of ETV (≥ 2 yrs to ≤ 6 yrs), (n=7, 3) | 8.07 (24) | 16.03 (8)
  Cmax of ETV (> 6 yrs to ≤ 12 yrs), (n=9, 7) | 6.29 (25) | 19.01 (15)
  Cmax of ETV (> 12 yrs to ≤ 18 yrs), (n=8,9) | 5.11 (27) | 11.32 (37)
  Cmin of ETV (≥ 2 yrs to ≤ 6 yrs), (n=7, 3) | 0.244 (32) | 0.468 (17)
  Cmin of ETV (> 6 yrs to ≤ 12 yrs), (n=9, 7) | 0.320 (22) | 0.497 (32)
  Cmin of ETV (> 12 yrs to ≤ 18 yrs), (n=8,9) | 0.271 (25) | 0.455 (25)

2. Secondary Outcome: Median Time of Maximum Observed Plasma Concentration (Tmax) in LVD-naive and LVD-experienced Participants, by Age Cohort
Description: Tmax was derived from plasma concentration of ETV versus time and measured in hours (h). Blood samples were obtained before study drug administration and at 0.5, 1, 2, 4, 8, and 24 hours after study drug administration on Day 14 (+/- 4 days) for the PK assessment. Plasma samples were analyzed for ETV with a validated method using liquid chromatography-tandem mass spectrometry detection. Age categories presented below: participants age as of first day of dosing. PK assessment was optional for Group C participants (NA-experienced participants who were included with the September 2011 country-specific protocol amendment). No Group C participants chose to participate in the PK assessment.
Time Frame: Day 14
Population: Participants in Groups A and B who received study drug and had PK assessment.
Measure: Median (Full Range); unit: h
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B)
Number analyzed (Participants) | 24 | 19
h
  Tmax of ETV (≥ 2 yrs to ≤ 6 yrs), (n=7, 3) | 0.50 [0.5 to 1.0] | 1.00 [0.5 to 1.5]
  Tmax of ETV (> 6 yrs to ≤ 12 yrs), (n=9, 7) | 0.57 [0.5 to 2.0] | 0.72 [0.5 to 1.0]
  Tmax of ETV (> 12 yrs to ≤ 18 yrs), (n=8,9) | 0.78 [0.5 to 1.0] | 0.52 [0.5 to 1.0]

3. Secondary Outcome: Mean Area Under the Concentration-Time Curve in One Dosing Interval [AUC(TAU)] of Entecavir in LVD-naive and LVD-experienced Participants, by Age Cohort
Description: Area under the Curve (AUC) was derived from plasma concentration of ETV versus time. AUC(TAU) was calculated by log- and linear trapezoidal summations, TAU = 24 hours, and was measured in nanograms*hours per milliliter (ng*h/mL). Blood samples were obtained before study drug administration and at 0.5, 1, 2, 4, 8, and 24 hours after study drug administration on Day 14 (+/- 4 days) for the PK assessment. Plasma samples were analyzed for ETV with a validated method using liquid chromatography-tandem mass spectrometry detection. PK assessment was optional for Group C participants (NA-experienced participants who were included with the September 2011 country-specific protocol amendment). No Group C participants chose to participate in the PK assessment.
Time Frame: Day 14
Population: Participants in Groups A and B who received study drug and had PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Lamivudine (LVD)-Naive (Group A): Participants with < 1 week of prior LVD therapy and with no LVD therapy within 24 weeks prior to enrollment were included in Group A. Prior to PK assessment, Cohort 1 (age ≥ 2 years to ≤ 6 years) and Cohort 2 (>6 years to ≤ 12 years) received ETV oral solution, 0.015 mg/kg up to 0.5 mg, once a day (QD) and Cohort 3 (age >12 years to ≤18 years) received ETV oral solution, 0.015 mg/kg up to 0.5 mg, or ETV tablets, 0.5 mg, QD. Following PK analysis, those who met the specified dosing requirements (at least 0.5 mg/day) and could tolerate swallowing ETV tablets were allowed to choose either formulation. Entecavir (ETV) was administered for a maximum of 120 weeks.
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B)
Number analyzed (Participants) | 24 | 19
ng*h/mL
  AUC(TAU) of ETV (≥ 2 yrs to ≤ 6 yrs), (n=7, 3) | 18.69 (21) | 42.26 (27)
  AUC(TAU) of ETV (> 6 yrs to ≤ 12 yrs), (n=9, 7) | 20.42 (20) | 41.50 (21)
  AUC(TAU) of ETV (> 12 yrs to ≤ 18 yrs), (n=8,9) | 15.96 (22) | 35.36 (24)

4. Secondary Outcome: Mean Apparent Total Body Clearance (CLT/F) of Entecavir in LVD-naive and LVD-experienced Participants, by Age Cohort
Description: CLT/F was calculated by dividing the dose of ETV by AUC(TAU) of ETV and was measured in liters per hour (L/h). Blood samples were obtained before study drug administration and at 0.5, 1, 2, 4, 8, and 24 hours after study drug administration on Day 14 (+/- 4 days) for the PK assessment. Plasma samples were analyzed for ETV with a validated method using liquid chromatography-tandem mass spectrometry detection. PK assessment was optional for Group C participants (NA-experienced participants who were included with the September 2011 country-specific protocol amendment). No Group C participants chose to participate in the PK assessment.
Time Frame: At 2 weeks
Population: Participants in Groups A and B who received study drug and had PK assessment.
Measure: Mean (Standard Deviation); unit: L/h
Groups:
- Lamivudine (LVD)-Experienced (Group B): Participants with > 12 weeks of prior LVD therapy were included in Group B. Prior to PK assessment, Cohort 1 (age ≥ 2 years to ≤ 6 years) and Cohort 2 (> 6 years to ≤ 12 years) received ETV oral solution, 0.030 mg/kg up to 1.0 mg, QD and Cohort 3 (age >12 years to ≤18 years) received ETV oral solution, 0.030 mg/kg up to 1.0 mg, or ETV tablets, 1.0 mg QD. Following PK analysis, those who met the specified dosing requirements (at least 1.0 mg/day) and could tolerate swallowing ETV tablets were allowed to choose either formulation. Entecavir (ETV) was administered for a maximum of 120 weeks.
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B)
Number analyzed (Participants) | 24 | 19
L/h
  CLT/F of ETV (≥ 2 yrs to ≤ 6 yrs), (n=7, 3) | 11.40 (2.564) | 12.31 (3.102)
  CLT/F of ETV (> 6 yrs to ≤ 12 yrs), (n=9, 7) | 22.66 (6.134) | 21.67 (6.940)
  CLT/F of ETV (> 12 yrs to ≤ 18 yrs), (n=8,9) | 31.92 (6.429) | 28.95 (6.496)

5. Secondary Outcome: Number of Participants With HBV DNA Less Than 50 IU/mL Through Week 96 in Treated Participants
Description: Hepatitis B virus DNA by polymerase chain reaction (PCR) was measured using the Roche COBAS TaqMan - high pure system (HPS) assay and was reported in international units per milliliter (IU/mL). Baseline was the last value measured prior to or on the date of the first dose of study therapy.
Time Frame: Baseline to Week 96
Population: The intent-to-treat method of Non-Completer = Failure was used through Week 48 in which all treated participants were analyzed, and participants with missing data at the analysis week were considered failures. After Week 48, the method of Non-Completer = Missing was used, in which participants with missing data at the analysis week were excluded.
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Baseline | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 22 | 17 | 5
  Week 12 | 1 | 0 | 0
  Week 24: number analyzed (Participants) | 24 | 18 | 5
  Week 24 | 10 | 3 | 0
  Week 36: number analyzed (Participants) | 21 | 19 | 5
  Week 36 | 11 | 6 | 0
  Week 48: number analyzed (Participants) | 22 | 18 | 5
  Week 48 | 14 | 9 | 0
  Week 96: number analyzed (Participants) | 12 | 13 | 4
  Week 96 | 8 | 11 | 2

6. Secondary Outcome: Number of Participants With Hepatitis B e Antigen (HBeAg) Loss Through Week 96 in Treated Participants
Description: HBeAg loss: HBeAg negative. The method used for the detection of HBe Ag was the DiaSorin - Anti HBe enzyme immunoassay kit. Baseline was the last value measured prior to or on the date of the first dose of study therapy.
Time Frame: Baseline to Week 96
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Baseline | 0 | 0 | 0
  Week 12 | 3 | 0 | 0
  Week 24 | 4 | 1 | 0
  Week 36: number analyzed (Participants) | 23 | 19 | 5
  Week 36 | 5 | 1 | 0
  Week 48 | 10 | 3 | 0
  Week 96: number analyzed (Participants) | 12 | 13 | 4
  Week 96 | 5 | 2 | 0

7. Secondary Outcome: Number of Participants With Hepatitis B s Antigen (HBsAg) Loss Through Week 96 in Treated Participants
Description: HBsAg loss: HBsAg negative. The method used for detection of HBsAg was the ADVIA Centaur iImmunoassay system. Baseline was the last value measured prior to or on the date of the first dose of study therapy.
Time Frame: Baseline to Week 96
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Baseline | 0 | 0 | 0
  Week 12 | 0 | 0 | 0
  Week 24 | 0 | 0 | 0
  Week 36 | 1 | 0 | 0
  Week 48 | 1 | 0 | 0
  Week 96: number analyzed (Participants) | 12 | 13 | 4
  Week 96 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Hepatitis B e Antigen Seroconversion Through Week 96 in Treated Participants
Description: HBe seroconversion: loss of HBeAg (HBeAg negative) with positive HB e antibodies (HBeAb), ie both the presence of HBeAb and the absence of HBeAg. The method used for the detection HBeAg seroconversion was the DiaSorin - Anti HBe enzyme immunoassay kit. Baseline was the last value measured prior to or on the date of the first dose of study therapy.
Time Frame: Baseline through Week 96
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Baseline | 0 | 0 | 0
  Week 12 | 3 | 0 | 0
  Week 24 | 4 | 1 | 0
  Week 36: number analyzed (Participants) | 23 | 19 | 5
  Week 36 | 5 | 1 | 0
  Week 48 | 10 | 3 | 0
  Week 96: number analyzed (Participants) | 12 | 13 | 4
  Week 96 | 5 | 1 | 0

9. Primary Outcome: Number of Participants With Serious Adverse Events (SAE) and Discontinuations Due to Adverse Events (AEs) - On Treatment
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Medical Dictionary for Regulatory Activities (MedDRA) version 16.0 was used.
Time Frame: Day 1 to Week 120
Population: All participants who received at least one dose of study drug. On-treatment period began on the first day of study therapy and ended 5 days after the last dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Serious Adverse Events (n=24, 19, 5) | 2 | 0 | 0
  Discontinuations Due to AEs (n=24,19,5) | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With HBV DNA Less Than Lower Limit of Detection (LLD) for the Roche COBAS TaqMan - HPS Assay at Week 96 in Treated Participants
Description: Hepatitis B virus DNA by PCR was measured using the Roche COBAS TaqMan - HPS assay and was reported in IU/mL. LLD = 6 IU/mL). Baseline was the last value measured prior to or on the date of the first dose of study therapy.
Time Frame: Baseline to Week 96
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Baseline | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 22 | 17 | 5
  Week 12 | 1 | 0 | 0
  Week 24: number analyzed (Participants) | 24 | 18 | 5
  Week 24 | 6 | 1 | 0
  Week 36: number analyzed (Participants) | 21 | 19 | 5
  Week 36 | 7 | 5 | 0
  Week 48: number analyzed (Participants) | 22 | 18 | 5
  Week 48 | 13 | 6 | 0
  Week 96: number analyzed (Participants) | 12 | 13 | 4
  Week 96 | 8 | 8 | 1

11. Secondary Outcome: Number of Participants With HBV DNA Less Than Lower Limit of Quantification (LLQ) for the Roche COBAS TaqMan - HPS Assay Through Week 96 in Treated Participants
Description: Hepatitis B virus DNA by PCR was measured using the Roche COBAS TaqMan - HPS assay and was reported in IU/mL. LLQ = 29 IU/mL. Baseline was the last value measured prior to or on the date of the first dose of study therapy.
Time Frame: Baseline through Week 96
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Baseline | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 22 | 17 | 5
  Week 12 | 1 | 0 | 0
  Week 24: number analyzed (Participants) | 24 | 18 | 5
  Week 24 | 9 | 2 | 0
  Week 36: number analyzed (Participants) | 21 | 19 | 5
  Week 36 | 10 | 5 | 0
  Week 48: number analyzed (Participants) | 22 | 18 | 5
  Week 48 | 14 | 7 | 0
  Week 96: number analyzed (Participants) | 12 | 13 | 4
  Week 96 | 8 | 8 | 2

12. Secondary Outcome: Number of Participants With HB s Antigen (HBsAg) Seroconversion Through Week 96 in Treated Participants
Description: HB s Ag seroconversion: loss of HBsAg (HBsAg negative) and presence of HB s antibodies (HBsAb). The method used for the detection of HBsAg seroconversion was the ADVIA Centaur iImmunoassay system. Baseline was the last value measured prior to or on the date of the first dose of study therapy.
Time Frame: Baseline through Week 96
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Baseline | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 20 | 19 | 5
  Week 12 | 0 | 0 | 0
  Week 24 | 0 | 0 | 0
  Week 36 | 0 | 0 | 0
  Week 48 | 0 | 0 | 0
  Week 96: number analyzed (Participants) | 12 | 13 | 4
  Week 96 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants Who Had a Protocol Defined Response (PDR) Through Week 96 in Treated Participants
Description: PDR was defined as confirmed HBV DNA < 50 IU/mL plus confirmed HBeAg seroconversion on 2 sequential measurements at least 14 days apart. Baseline was the last value measured prior to or on the date of the first dose of study therapy.
Time Frame: Baseline to Week 96
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Week 12 | 0 | 0 | 0
  Week 24 | 4 | 0 | 0
  Week 36 | 4 | 1 | 0
  Week 48 | 7 | 3 | 0
  Week 96: number analyzed (Participants) | 12 | 13 | 4
  Week 96 | 3 | 1 | 0

14. Secondary Outcome: Mean Log10 Change From Baseline in HBV DNA Using Roche COBAS TaqMan - HPS Through Week 96 in Treated Participants
Description: Hepatitis B virus DNA by PCR was measured using the Roche COBAS TaqMan - HPS assay and was reported in IU/mL. HBV DNA log10 changes from baseline were summarized over time.
Time Frame: Baseline to Week 96
Population: Participants who received at least one dose of study drug, and had a measurement at baseline and at the specific analysis week.
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
IU/mL
  Week 12: number analyzed (Participants) | 22 | 17 | 5
  Week 12 | -4.45 (0.2418) | -3.89 (0.1592) | -3.80 (0.4657)
  Week 24: number analyzed (Participants) | 24 | 18 | 5
  Week 24 | -5.30 (0.2744) | -4.85 (0.2900) | -3.89 (0.5440)
  Week 36: number analyzed (Participants) | 21 | 19 | 5
  Week 36 | -5.61 (0.2580) | -5.14 (0.2604) | -3.90 (0.2499)
  Week 48: number analyzed (Participants) | 22 | 18 | 5
  Week 48 | -5.86 (0.2176) | -5.36 (0.3032) | -4.32 (0.4794)
  Week 96: number analyzed (Participants) | 12 | 13 | 4
  Week 96 | -6.30 (0.2576) | -5.86 (0.2222) | -5.79 (0.5308)

15. Secondary Outcome: Alanine Aminotransferase (ALT) Normalization From Baseline Through Week 96 in Treated Participants
Description: Normalization in ALT= ALT ≤ 1.0*upper limit of normal (ULN). Baseline was the last value measured prior to or on the date of the first dose of study therapy.
Time Frame: Baseline to Week 96
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Baseline | 0 | 1 | 2
  Week 4 | 1 | 1 | 2
  Week 8 | 3 | 2 | 2
  Week 12 | 5 | 7 | 3
  Week 18 | 15 | 10 | 5
  Week 24 | 15 | 12 | 5
  Week 30 | 16 | 13 | 5
  Week 36 | 16 | 16 | 5
  Week 42 | 16 | 15 | 5
  Week 48 | 20 | 18 | 4
  Week 96: number analyzed (Participants) | 11 | 13 | 4
  Week 96 | 10 | 13 | 3

16. Secondary Outcome: Number of Participants With HBV DNA by PCR Categories at Weeks 48 and 96 in Treated Participants
Description: as for outcome 11
Time Frame: Baseline, Week 48, Week 96
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Baseline >=17,200 IU/mL | 24 | 19 | 5
  Week 48: < 50 IU/mL: number analyzed (Participants) | 22 | 19 | 5
  Week 48: < 50 IU/mL | 14 | 9 | 0
  Week 48: 50 - < 172 IU/mL: number analyzed (Participants) | 22 | 19 | 5
  Week 48: 50 - < 172 IU/mL | 1 | 2 | 0
  Week 48: 172 - < 1720 IU/mL: number analyzed (Participants) | 22 | 19 | 5
  Week 48: 172 - < 1720 IU/mL | 3 | 3 | 1
  Week 48: 1720 - < 17,200 IU/mL: number analyzed (Participants) | 22 | 19 | 5
  Week 48: 1720 - < 17,200 IU/mL | 3 | 1 | 3
  Week 48: > = 17,200 IU/mL: number analyzed (Participants) | 22 | 19 | 5
  Week 48: > = 17,200 IU/mL | 1 | 3 | 1
  Week 96: < 50 IU/mL: number analyzed (Participants) | 12 | 13 | 4
  Week 96: < 50 IU/mL | 8 | 11 | 2
  Week 96: 50 - < 172 IU/mL: number analyzed (Participants) | 12 | 13 | 4
  Week 96: 50 - < 172 IU/mL | 1 | 1 | 0
  Week 96: 172 - < 1720 IU/mL: number analyzed (Participants) | 12 | 13 | 4
  Week 96: 172 - < 1720 IU/mL | 3 | 0 | 1
  Week 96: 1720 - < 17,200 IU/mL: number analyzed (Participants) | 12 | 13 | 4
  Week 96: 1720 - < 17,200 IU/mL | 0 | 1 | 1
  Week 96: > = 17,200 IU/mL: number analyzed (Participants) | 12 | 13 | 4
  Week 96: > = 17,200 IU/mL | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With a Combination of ALT Normalization and HBV DNA Less Than 50 IU/mL Through Week 96 in Treated Participants
Description: Hepatitis B virus DNA by PCR was measured using the Roche COBAS TaqMan - HPS assay and was reported in IU/mL. Baseline was the last value measured prior to or on the date of the first dose of study therapy. Normalization in ALT= ALT ≤ 1.0*ULN.
Time Frame: Baseline to Week 96
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Baseline | 0 | 0 | 0
  Week 12 | 0 | 0 | 0
  Week 24 | 10 | 3 | 0
  Week 36 | 11 | 4 | 0
  Week 48 | 13 | 9 | 0
  Week 96 | 7 | 11 | 2

18. Secondary Outcome: Number of Participants With a Combination of ALT Normalization and HBV DNA Less Than 50 IU/mL, Plus HBeAg Seroconversion Through Week 96 in Treated Participants
Description: Hepatitis B virus DNA by PCR was measured using the Roche COBAS TaqMan - HPS assay and was reported in IU/mL. Baseline was the last value measured prior to or on the date of the first dose of study therapy. Normalization in ALT= ALT ≤ 1.0*ULN. HBe seroconversion was determination of presence of HBeAb and loss of HBeAg. The method used for the detection of HBeAg seroconversion was the DiaSorin - Anti HBe enzyme immunoassay kit.
Time Frame: Baseline to Week 96
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Baseline | 0 | 0 | 0
  Week 12 | 0 | 0 | 0
  Week 24 | 4 | 0 | 0
  Week 36: number analyzed (Participants) | 22 | 19 | 5
  Week 36 | 4 | 1 | 0
  Week 48: number analyzed (Participants) | 23 | 19 | 5
  Week 48 | 8 | 3 | 0
  Week 96: number analyzed (Participants) | 11 | 13 | 4
  Week 96 | 3 | 1 | 0

19. Secondary Outcome: Number of Participants With a Combination of ALT Normalization and HBV DNA Less Than 50 IU/mL, Without HBeAg Seroconversion, Through Week 96 in Treated Participants
Description: Hepatitis B virus DNA by PCR was measured using the Roche COBAS TaqMan - HPS assay and was reported in IU/mL. Baseline was the last value measured prior to or on the date of the first dose of study therapy. Normalization in ALT= ALT ≤ 1.0*ULN. HBe seroconversion: loss of HBeAg (HBeAg negative) with positive HBeAb. The method used for the detection of HBeAg/Ab serologies was the DiaSorin enzyme immunoassay kit.
Time Frame: Baseline to Week 96
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Baseline | 0 | 0 | 0
  Week 12 | 0 | 0 | 0
  Week 24 | 6 | 3 | 0
  Week 36: number analyzed (Participants) | 23 | 19 | 5
  Week 36 | 7 | 3 | 0
  Week 48 | 5 | 6 | 0
  Week 96: number analyzed (Participants) | 12 | 13 | 4
  Week 96 | 4 | 10 | 2

20. Secondary Outcome: Number of Participants With Hematology Laboratory Abnormalities (Grades 1 - 4) - On Treatment - Treated Participants
Description: Toxicity Scale: Division of AIDs (DAIDS) grades Version 1.0. Upper limit of normal (ULN); lower limit of normal (LLN); Cells per Liter (c/L); cells per microliter (c/µL); grams per deciliter (g/dL); milliequivalents per liter (mEq/L); cells per microliter (c/µL): Grade (Gr). Hemoglobin g/dL: Gr1:10.0-10.9;Gr2: 9.0-9.9; Gr3:7.0-8.9; Gr4: <7.0. International normalization ratio (INR): Gr1:1.1-<1.5*ULN; Gr2: 1.6-<2.0*ULN; Gr3: 2.1-3.0*ULN;Gr4: >3.0*ULN. Neutrophils/bands c/µL: Gr1;1.0-1.3*10^3; Gr2: 0.75-0.99*10^3; Gr 3: 0.50-0.749*10^3; Gr4: <0.5*10^3.
Time Frame: Day 1 to Week 120
Population: Participants who received at least 1 dose of study therapy, and had a measurement during the on-treatment period (i.e., after the first day of study therapy through 5 days after the last dose of study therapy).
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Hemoglobin | 1 | 0 | 1
  International normalization ratio | 4 | 3 | 0
  Neutrophils (absolute) + bands | 3 | 3 | 0

21. Secondary Outcome: Number of Participants With Chemistry Laboratory Abnormalities (Grades 1 - 4) - On Treatment - Treated Participants
Description: Toxicity Scale: DAIDS Version 1.0 and modified World Health Organization (WHO). Grade (Gr). ALT: Gr1:1.25-<2.5*ULN; Gr2: 2.6-<5.0 *ULN; Gr3: 5.1-10.0*ULN; Gr4:>10.0*ULN. Aspartate aminotransferase (AST): Gr1: 1.25-<2.5*ULN; Gr2:2.6-<5.0*ULN; Gr 3: 5.1-10.0*ULN; Gr4>10.0*ULN. Alkaline phosphatase: Gr1:1.25-<2.5*ULN; Gr2: 2.6-<5.0*ULN; Gr3: 5.1-10.0*ULN; Gr4: >10.0*ULN. Lipase: Gr1:1.1-<1.5*ULN;Gr2:1.6-<3.0*ULN; Gr3: 3.1-5.0*ULN; Gr4: >5.0*ULN. Creatinine: Gr1: 1.1-1.3*ULN; Gr2: 1.4-<1.8*ULN; Gr3: 1.9 - <3.4*ULN; Gr4: >=3.5*ULN. Glucose mg/dL (high): Gr1:110-<125 (Fasting)/116-<160;Gr2:126-<250 (F)/161-<250; Gr3: 251-500; Gr4: >500.Glucose (low): Gr1: 55-64; Gr2: 40 - <54; Gr3: 30-39; Gr4: <30 mg/dL.
Time Frame: Day 1 to Week 120
Population: Participants who received at least one dose of study drug, and had a measurement during the on-treatment period (i.e., after the first day of study therapy through 5 days after the last dose of study therapy).
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  ALT | 23 | 17 | 4
  AST | 14 | 9 | 1
  Alkaline Phosphatase | 3 | 3 | 0
  Lipase | 5 | 12 | 3
  Creatinine | 1 | 1 | 0
  Glucose, high | 3 | 4 | 1
  Glucose, low | 3 | 4 | 1

22. Secondary Outcome: Number of Participants With Electrolyte Laboratory Abnormalities (Grades 1 - 4) - On Treatment - Treated Participants
Description: Toxicity Scale: DAIDS Version 1.0 and modified World Health Organization (WHO) for chloride. Milliequivalents per liter (mEq/L); Grade (Gr). Chloride high (mEq/L): Gr1: 113-<117; Gr2: 117-<121; Gr3: 121-125; Gr4: >125. Potassium low (mEq/L): Gr1: 3.0-3.4; Gr2: 2.5-2.9; Gr3:2.0-<2.4; Gr4: <2.0. Potassium high: Gr1; 5.6- <6.0; Gr2: 6.1-<6.5; Gr3: 6.6-7.0; Gr4: >7.0. Sodium high (mEq/L): Gr1; 146-<150; Gr2: 151-<154; Gr3: 155-<159; Gr4: >=160.
Time Frame: Day 1 Week 120
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Lamivudine (LVD)-Naive (Group A) | Lamivudine (LVD)-Experienced (Group B) | Nucleoside/Tide Analog (NA) - Experienced (Group C)
Number analyzed (Participants) | 24 | 19 | 5
participants
  Chloride, high | 3 | 0 | 0
  Potassium, low | 1 | 0 | 0
  Potassium, high | 1 | 1 | 0
  Sodium, high | 4 | 3 | 0

ADVERSE EVENTS:
Time Frame: From first dose to date of last dose plus 5 days, up to 120 weeks
Groups:
- Group A LVD-naive: Participants with < 1 week of prior LVD therapy and with no LVD therapy within 24 weeks prior to enrollment were included in Group A. Prior to PK assessment, Cohort 1 (age ≥ 2 years to ≤ 6 years) and Cohort 2 (>6 years to ≤ 12 years) received ETV oral solution, 0.015 mg/kg up to 0.5 mg, once a day (QD) and Cohort 3 (age >12 years to ≤18 years) received ETV oral solution, 0.015 mg/kg up to 0.5 mg, or ETV tablets, 0.5 mg, QD. Following PK analysis, those who met the specified dosing requirements (at least 0.5 mg/day) and could tolerate swallowing ETV tablets were allowed to choose either formulation. Entecavir (ETV) was administered for a maximum of 120 weeks.
- Group B LVD-exp: Participants with > 12 weeks of prior LVD therapy were included in Group B. Prior to PK assessment, Cohort 1 (age ≥ 2 years to ≤ 6 years) and Cohort 2 (> 6 years to ≤ 12 years) received ETV oral solution, 0.030 mg/kg up to 1.0 mg, QD and Cohort 3 (age >12 years to ≤18 years) received ETV oral solution, 0.030 mg/kg up to 1.0 mg, or ETV tablets, 1.0 mg QD. Following PK analysis, those who met the specified dosing requirements (at least 1.0 mg/day) and could tolerate swallowing ETV tablets were allowed to choose either formulation. Entecavir (ETV) was administered for a maximum of 120 weeks.
- Group C NA-exp: Participants who failed previous treatment with any non-ETV nucleoside/tide analog (NA) were included in Group C, starting in 2011. PK assessment was optional to participants in Group C. All participants received ETV oral solution, 0.030 mg/kg up to 1.0 mg, or ETV tablets, 1.0 mg, QD. Participants who met the specified dosing requirements (at least 1.0 mg/day for NA-experienced participants) and could tolerate swallowing ETV tablets were allowed to choose either formulation. ETV was administered for a maximum of 120 weeks.
Arm/Group | Group A LVD-naive | Group B LVD-exp | Group C NA-exp
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/19 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/24 | 0/19 | 0/5
Other Adverse Events (participants affected / at risk) | 21/24 | 17/19 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A LVD-naive (N=24) | Group B LVD-exp (N=19) | Group C NA-exp (N=5)
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A LVD-naive (N=24) | Group B LVD-exp (N=19) | Group C NA-exp (N=5)
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 1
Enteritis (Gastrointestinal disorders) | 1 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 1
Chest pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 0
Influenza like illness (General disorders) | 1 | 2 | 0
Pyrexia (General disorders) | 10 | 5 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Impetigo (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 0
Lyme disease (Infections and infestations) | 0 | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 1
Mumps (Infections and infestations) | 0 | 1 | 0
Otitis externa (Infections and infestations) | 2 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 3 | 2
Viral upper respiratory tract infection (Infections and infestations) | 4 | 9 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 7 | 5 | 0
Product taste abnormal (Product Issues) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.